CLINICAL TRIAL: NCT02731092
Title: Safety and Tolerability of Lactoferrin in Very Low Birth Weight Infants
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Collaborators: The Gerber Foundation (Other)
Responsible Party: Principal Investigator, David A Kaufman, MD, University of Virginia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-HSR 18130
Record Dates: First submitted 2016-03-18; First posted 2016-04-07 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Very Low Birth Weight Infants
Keywords: lactoferrin; very low birth weight infants; preterm infants
MeSH Terms: interventions — Lactoferrin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Lactoferrin 100 mg/kg (Experimental): 100 mg/kg enteral administration daily for 30 days
  Interventions: Dietary Supplement: Lactoferrin
- Lactoferrin 200 mg/kg (Experimental): 200 mg/kg enteral administration daily for 30 days
  Interventions: Dietary Supplement: Lactoferrin
- Lactoferrin 300 mg/kg (Experimental): 300 mg/kg enteral administration daily for 30 days
  Interventions: Dietary Supplement: Lactoferrin

INTERVENTIONS:
Dietary Supplement: Lactoferrin — Bovine Lactoferrin 100 mg/ml dissolved in sterile water
  Other Names: Bioferrin® 2000

SUMMARY:
To evaluate the safety and tolerability of three different lactoferrin doses in preterm infants

DETAILED DESCRIPTION:
Aim1: To evaluate the safety and tolerability of three different lactoferrin doses in preterm infants

1. Lactoferrin related adverse events and serious adverse events
2. Number of infants reaching full feeds while receiving lactoferrin (120 ml/kg/day)
3. Episodes of not receiving enteral feedings for > 24 hours once feeding is initiated

Aim 2: To evaluate lactoferrin absorption and excretion.

1. Examine lactoferrin levels in saliva, urine, plasma and stool
2. Examine lactoferrin levels in maternal and human donor milk.

Aim 3: To evaluate the effect of lactoferrin on the intestinal microbiome structure.

ELIGIBILITY:
Inclusion Criteria:

* < 15 days of age and receiving enteral feedings
* < 1500 grams birth weight
* <37 weeks gestation

Exclusion Criteria:

* Congenital bowel obstruction ( esophageal, duodenal, small bowel or anal atresias, Hirschsprung disease, malrotation)
* Known necrotizing enterocolitis or bowel perforation

Max Age: 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2016-04; Primary Completion 2016-12 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Definitely related study solution serious adverse event | 30 days while receiving study solution

SECONDARY OUTCOMES:
Number of infants reaching 120 ml/kg of enteral feeds | 30 days while receiving study solution
  Number of infants reaching 120 ml/kg of enteral feeds while receiving study solution
Number of days not receiving any feedings after lactoferrin administration | 30 days while receiving study solution
  Number of days not receiving any feedings after lactoferrin administration begun

CONTACTS AND LOCATIONS:
Overall Officials: David A Kaufman, MD, Principal Investigator — University of Virginia School of Medicine
Locations (2):
- United States (2):
  - University of Virginia Neonatal Intensive Care Unit, Charlottesville, Virginia
  - University of Virginia HealthSystem, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
At UVA and MTA with outside institutions